CLINICAL TRIAL: NCT02080858
Title: The Effect of Ticagrelor and Apixaban With or Without Acetylsalicylic Acid on Markers of Coagulation Activation at the Site of Thrombus Formation in Vivo in Healthy Male Subjects and in an ex Vivo Perfusion Chamber Model at High and Low Shear Rate
Brief Title: Triple vs. Dual Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wolzt, Prof. MD, Prof. MD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TVDAT-1.0
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation; Acute Coronary Syndrome
Keywords: Apixaban; Ticagrelor; ASA; shed blood; perfusion chamber
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome | interventions — Ticagrelor; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor + Apixaban + ASA (Experimental): 180 mg Ticagrelor loading dose + apixaban 2.5 mg bid + 300 mg ASA loading dose (day 1) followed by ticagrelor 90 mg bid + apixaban 2.5 mg + 100 mg ASA od to reach steady state conditions within 4.5 days
  Interventions: Drug: Ticagrelor + Apixaban + ASA
- Ticagrelor + Apixaban (Active Comparator): 180mg ticagrelor loading dose + apixaban 2.5 mg bid (day 1) followed by ticagrelor 90 mg bid + apixaban 2.5 mg to reach steady state conditions within 4.5 days
  Interventions: Drug: Ticagrelor + Apixaban

INTERVENTIONS:
Drug: Ticagrelor + Apixaban + ASA
  Arms: Ticagrelor + Apixaban + ASA
Drug: Ticagrelor + Apixaban
  Arms: Ticagrelor + Apixaban

SUMMARY:
Background:

The acute coronary syndrome (ACS) is a complication of coronary artery disease (CAD) and associated with increased mortality. Dual antiplatelet therapy of acetylsalicylic acid (ASA) with P2Y12 receptor antagonists such as clopidogrel is a cornerstone in the treatment of patients with advanced CAD. Due to delayed onset of action, intersubject variability or resistance to clopidogrel, different platelet aggregation inhibitors have been developed. Ticagrelor is a reversible P2Y12 receptor antagonist with superior efficacy compared to clopidogrel in the prevention of cardiovascular death in these patients.

Atrial fibrillation (AF) is also associated with thromboembolic events and substantial mortality. Beside vitamin K antagonists (VKA, phenprocoumon) for stroke prevention in patients with AF, the direct factor Xa inhibitor apixaban has recently received approval for prophylactic treatment of patients with non-valvular AF.

However, there is a lack of efficacy or safety data for the combined impact of antithrombotic drugs in patients requiring arterial and venous thromboembolic prophylaxis due to their underlying co-morbidities. One trial suggests treatment with VKA + clopidogrel without ASA as equal effective as antithrombotic triple therapy (with ASA) in this population. However, the effect in combination with novel oral anticoagulants has not been investigated so far.

Study objectives:

To evaluate the effect of ticagrelor + apixaban in combination with or without ASA at steady state on markers of coagulation activation and on thrombus size in an ex vivo perfusion chamber experiment. Additionally, plasma samples will be analysed for PK-data (ticagrelor & apixaban concentrations)

Study design:

A single-centre, prospective, sequential, controlled, analyst-blinded study in two groups. Subjects will receive ticagrelor + apixaban in combination with (study A) or without (study B) ASA. All IMPs will be administered at doses indicated for stroke prevention in AF (lower dose: 2.5mg due to ethical concerns) or ACS. Markers on thrombin generation and platelet activation will be studied in venous blood where coagulation is in resting state and in shed blood where the clotting system is activated in the microvasculature in vivo: prothrombin fragment 1+2 (F1+2), thrombin-anti-thrombin (TAT), β-thromboglobulin (β-TG). Additionally, inhibition of factor Xa activity and concentrations of ticagrelor and apixaban will be assessed in venous blood. Further, thrombus size of clots formed in an ex vivo perfusion chamber will be determined by measurement of D-Dimer and p-Selectin levels.

Study population A total of 40 healthy, non-smoking and drug-free male volunteers will be enrolled (study A and B; n = 20 per group).

Main outcome variables:

* β-TG in shed blood

Additional outcome variables:

* F1+2 and TAT in shed blood
* fibrin formation (D-Dimer) and platelet deposition (p-Selectin) in an ex vivo perfusion chamber model of thrombosis
* β-TG, F1+2, TAT & inhibition of factor Xa in venous blood
* PT, aPTT and ACT in venous blood
* ticagrelor & apixaban plasma concentrations
* shed blood volume

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects; 18 - 40 years of age
* body mass index between 18 and 27 kg/m2
* Written informed consent
* Normal findings in medical & bleeding history
* Non-smoking behaviour

Exclusion Criteria:

* Regular intake of any medication including OTC drugs and herbals within 2 weeks before IMP administration
* Known coagulation disorders (e.g. haemophilia, von Willebrand´s disease)
* Known disorders with increased bleeding risk (e.g. peridontitis, haemorrhoids, acute gastritis, peptic ulcer, intestinal ulcer)
* Known sensitivity to common causes of bleeding (e.g. nasal)
* History of thromboembolism
* Anaemia (defined as haemoglobin levels < LLN)
* Impaired liver function (AST, ALT, GGT >2 x ULN, Bilirubin >1.5 x ULN)
* Impaired renal function (serum creatinine > 1.3 mg/dl)
* Any other relevant deviation from the normal range in clinical chemistry, haematology or urine analysis
* HIV-1/2-Ab, HbsAg or HCV-Ab positive serology
* Systolic blood pressure above 145 mmHg, diastolic blood pressure above 95 mmHg
* Known allergy against test agents
* Regular daily consumption of more than on litre of xanthine-containing beverages or more than 40g alcohol
* Participation in another clinical trial during the preceding 3 weeks

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
β-thromboglobulin (β-TG) | Changes in shed blood from baseline, at 3 hours, at trough and peak steady state conditions
  Of primary interest is the difference in shed blood β-TG "3h post-dose at steady state (peak)" or "pre-dose at steady state (trough)" and Baseline during triple therapy vs. dual therapy.

SECONDARY OUTCOMES:
Prothrombin fragment F1+2 (F1+2) | Changes in shed blood from baseline, at 3 hours, at trough and peak steady state conditions
  Of primary interest is the difference in shed blood F1+2 "3h post-dose at steady state (peak)" or "pre-dose at steady state (trough)" and Baseline during triple therapy vs. dual therapy.
Thrombin-Anti-Thrombin (TAT) | Changes in shed blood from baseline, at 3 hours, at trough and peak steady state conditions
  Of primary interest is the difference of TAT in shed blood "3h post-dose at steady state (peak)" or "pre-dose at steady state (trough)" and Baseline during triple therapy vs. dual therapy.
D-dimer | Changes from baseline, at 3 hours, at trough and peak steady state conditions
  Changes on fibrin formation in an ex vivo perfusion chamber model of thrombosis at high and low shear rate. Of primary interest is the difference in D-Dimer "3h post-dose at steady state (peak)" or "pre-dose at steady state (trough)" and Baseline during triple therapy vs. dual therapy.
P-selectin | Changes from baseline, at 3 hours, at trough and peak steady state conditions
  Changes on platelet deposition in an ex vivo perfusion chamber model of thrombosis at high and low shear rate. Of primary interest is the difference in D-Dimer "3h post-dose at steady state (peak)" or "pre-dose at steady state (trough)" and Baseline during triple therapy vs. dual therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria